CLINICAL TRIAL: NCT00373113
Title: Phase III Randomized, Multi Center Study Of Sunitinib Malate (SU 011248) Or Capecitabine In Subjects With Advanced Breast Cancer Who Failed Both A Taxane And An Anthracycline Chemotherapy Regimen Or Failed With A Taxane And For Whom Further Anthracycline Therapy Is Not Indicated
Brief Title: A Clinical Trial Comparing Efficacy And Safety Of Sunitinib And Capecitabine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181107
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Breast Neoplasms
Keywords: advanced breast cancer; metastatic breast cancer; treatment resistant; treatment failure
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 1250 mg/m^2, twice daily, for 2 consecutive weeks, followed by a 1-week rest period and given as 3-week cycles
  Interventions: Drug: Capecitabine
- B (Experimental): 37.5 mg daily, continuous dosing
  Interventions: Drug: Sunitinib malate

INTERVENTIONS:
Drug: Capecitabine — 1250 mg/m^2, twice daily, for 2 consecutive weeks, followed by a 1-week rest period and given as 3-week cycles
  Other Names: xeloda
  Arms: A
Drug: Sunitinib malate — 37.5 mg daily, continuous dosing
  Other Names: sunitinib
  Arms: B

SUMMARY:
To compare efficacy and safety of Sunitinib and Capecitabine in subjects with advanced breast cancer who failed both a taxane and an anthracycline chemotherapy regimen or failed with a taxane and for whom further anthracycline therapy is not indicated

DETAILED DESCRIPTION:
Patient enrollment in this trial was discontinued based on statistical assessment for futility. An independent Data Monitoring Committee found that even if the trial had been allowed to continue, treatment with single agent sunitinib would be unable to demonstrate a statistically significant improvement in the primary endpoint of progression-free survival compared with single agent capecitabine in the study population. Pfizer notified clinical trial investigators involved in the study and regulatory agencies of these findings on 25Mar2009. Patients receiving sunitinib will be allowed to receive capecitabine or enter an extension trial if they are receiving clinical benefit from continued sunitinib therapy. There were no safety concerns leading to the decision to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* breast adenocarcinoma
* prior treatment with an anthracycline and a taxane either concurrently or sequentially in the neoadjuvant, adjuvant and or/ advanced disease treatment settings. No more than 1 chemotherapy regimen in the advanced setting

Exclusion Criteria:

* Prior treatment with regimens of chemotherapy in the advanced/metastatic disease setting beyond those containing anthracyclines and taxanes or multiple anthracyclines/ taxanes treatments.
* Any prior regimen with capecitabine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (111):
- Argentina (6):
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Bahía Blanca, Prov. de Buenos Aires
  - Pfizer Investigational Site, Viedma, Río Negro Province
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, San Miguel de Tucumán
- Australia (6):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Brazil (4):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (3):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
- Canada (4):
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Temuco, Región de la Araucanía, Chile
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogotá, Cundinamarca
- France (7):
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Neuilly-sur-Seine
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Rennes
- Germany (13):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, Leer
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Meiningen
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Offenburg
  - Pfizer Investigational Site, Tübingen
- Hong Kong (4):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Tuenmen
  - Pfizer Investigational Site, Wan Chai
- India (5):
  - Pfizer Investigational Site, Navrangpura / Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Italy (4):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Reggio Emilia
- Japan (9):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Kita-adachi-gun, Saitama
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chuo-Ku, Tokyo
- Mexico (7):
  - Pfizer Investigational Site, Chihuahua City, Chihuahua
  - Pfizer Investigational Site, Acapulco de Juárez, Guerrero
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, Puebla City, Puebla
  - Pfizer Investigational Site, Ciudad Obregón, Sonora
  - Pfizer Investigational Site, Toluca, State of Mexico
- Peru (2):
  - Pfizer Investigational Site, Lima, Lima Province
  - Pfizer Investigational Site, Lima
- Philippines (2):
  - Pfizer Investigational Site, Quezon City
  - Pfizer Investigational Site, San Juan City
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- South Africa (2):
  - Pfizer Investigational Site, Parktown
  - Pfizer Investigational Site, Sandton
- South Korea (5):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul
- Spain (13):
  - Pfizer Investigational Site, Mataró, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Jaén, Jaen
  - Pfizer Investigational Site, A Coruña, La Coruña
  - Pfizer Investigational Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Pfizer Investigational Site, Alcorcón, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Salamanca, Salamanca
  - Pfizer Investigational Site, Bilbao, Vizcaya
- Taiwan (5):
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
- United Kingdom (4):
  - Pfizer Investigational Site, Cardiff, South Wales
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Somerset

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181107&StudyName=A%20Clinical%20Trial%20Comparing%20Efficacy%20And%20Safety%20Of%20Sunitinib%20And%20Capecitabine

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: 37.5 milligrams (mg) daily, continuous dosing
- Capecitabine: 1250 milligrams per square meter (mg/m^2) or 1000 mg/m^2 in older participants, twice daily for 2 consecutive weeks, followed by a 1-week rest period and given as 3-week cycles
Period: Overall Study
Arm/Group | Sunitinib | Capecitabine
Started | 238 | 244
Received Treatment | 238 | 240
Completed | 0 | 0
Not Completed | 238 | 244
Not completed — Death | 1 | 7
Not completed — Adverse Event | 38 | 24
Not completed — Study terminated by sponsor | 9 | 1
Not completed — Global deterioration of health status | 10 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Objective progression or relapse | 150 | 169
Not completed — Other | 14 | 17
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib: 37.5 mg daily, continuous dosing
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Capecitabine | Total
Number analyzed (Participants) | 238 | 244 | 482
Age, Customized [Number; unit: Participants]
  18 to 44 years | 50 | 70 | 120
  45 to 64 years | 159 | 129 | 288
  > = 65 years | 29 | 45 | 74
Sex/Gender, Customized [Number; unit: Participants]
  Female | 238 | 244 | 482
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time from the date of randomization to the date of the first documentation of objective tumor progression or death due to any cause, whichever occured first.
Time Frame: From time of randomization to every 6 weeks thereafter through 22 months or until death
Population: Intent-to-treat (ITT) population: included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 238 | 244
Months | 2.8 [2.4 to 4.0] | 4.2 [3.8 to 5.5]
Statistical Analysis 1: Comparison: Sunitinib vs Capecitabine; Null hypothesis is that PFS (median=4.2 months) for sunitinib arm equals PFS for capecitabine arm. The study was designed to have 90% power to detect statistical difference in PFS between two treatment groups assuming the hazard ratio (sunitinib/capecitabine) is 0.75 and both arms follow exponential distribution; Test type: Superiority or Other; p = 0.002, Log Rank — 2-sided log-rank test with the same set of stratification factors. The set of stratification factors included those used in the randomization except study sites; Hazard Ratio (HR) = 1.470, 95% CI 2-sided [1.156 to 1.869] — Hazard ratio was calculated by the stratified Cox proportional hazards model

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time from randomization to first documentation of objective tumor progression.
Time Frame: From time of randomization to every 6 weeks thereafter through 22 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 238 | 244
Months | 2.8 [2.5 to 4.0] | 4.2 [3.8 to 5.5]
Statistical Analysis 1: Comparison: Sunitinib vs Capecitabine; Test type: Superiority or Other; p < 0.001, Log Rank — 2-sided log-rank test with the same set of stratification factors that was used in the randomization except study sites; Hazard Ratio (HR) = 1.516, 95% CI 2-sided [1.188 to 1.933] — Hazard ratio was calculated by the stratified Cox proportional hazards model

3. Secondary Outcome: Number of Participants With Overall Response (OR)
Description: OR was defined as the number of participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST, Version 1.0) for at least 4 weeks, confirmed by repeat tumor assessments. CR was defined as the disappearance of all target lesions. PR was defined as a greater than or equal to (>=) 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of randomization to every 6 weeks thereafter through 22 months
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 238 | 244
Participants | 27 | 40
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 11.3, 95% CI 2-sided [7.6 to 16.1]
Statistical Analysis 2: Comparison: Capecitabine; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 16.4, 95% CI 2-sided [12.0 to 21.6]
Statistical Analysis 3: Comparison: Sunitinib vs Capecitabine; Test type: Superiority or Other; p = 0.109, Pearson Chi-Square Test; Mean Difference (Final Values) = -5.049, 95% CI 2-sided [-11.2 to 1.1]

4. Secondary Outcome: Duration of Response (DR)
Description: Time from the first documentation of OR (CR or PR) that was subsequently confirmed to the first documentation of tumor progression or death due to any cause. CR was defined as disappearance of all target lesions. PR was defined as a >= 30% decrease in sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions.
Time Frame: From time of randomization to every 6 weeks thereafter through 22 months or death
Population: ITT population. DR was calculated for the subgroup of participants with objective response. 27 participants in the sunitinib arm and 40 participants in the capecitabine arm reported CR or PR response and were analyzed for DR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 27 | 40
Months | 6.9 [3.1 to 8.5] | 9.3 [5.5 to 9.7]
Statistical Analysis 1: Comparison: Sunitinib vs Capecitabine; Test type: Superiority or Other; p = 0.037, Log Rank; Hazard Ratio (HR) = 2.788, 95% CI 2-sided [1.042 to 7.459]

5. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time from randomization to the first documentation of objective tumor response (CR or PR) that was subsequently confirmed. CR was defined as disappearance of all target lesions. PR was defined as a >= 30% decrease in sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions.
Time Frame: From time of randomization to every 6 weeks thereafter through 22 months
Population: The study was stopped early for futility and TTR analysis was not performed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Average time from randomization to first documentation of death due to any cause.
Time Frame: From time of randomization until death
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 238 | 244
Months | 15.3 [12.0 to 24.7] | 16.9 [14.5 to 26.0]
Statistical Analysis 1: Comparison: Sunitinib vs Capecitabine; Test type: Superiority or Other; p = 0.219, Log Rank — 2-sided log-rank test with the same set of stratification factors that were used in the randomization except study sites; Hazard Ratio (HR) = 1.202, 95% CI 2-sided [0.896 to 1.611]

7. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 scales: functional (physical/role/cognitive/emotional/social), symptom (fatigue/nausea/vomiting/pain), global health/QOL, cancer symptom (dyspnea/insomnia/appetite loss/constipation/diarrhea).
  Feelings in past week: response range: not at all to very much, global/QOL range: very poor to excellent. Scales/single-items averaged, score 0 to 100. Higher functional/global=better functioning and symptom=greater degree of symptoms.
Time Frame: From Day 1 of Cycle 1, then odd numbered cycles thereafter
Population: The study was stopped early for futility and EORTC QLQ-C30 analysis was not performed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: EORTC QLQ Breast Cancer Module (BR23)
Description: BR23: measured disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm/shoulder pain, breast pain, swollen breast, and skin problems on the breast. Recall period: past week; response range: not at all to very much.
  Scale score range: 0 to 100. Higher symptom score implied a greater degree of symptoms.
Time Frame: From Day 1 of Cycle 1, then odd numbered cycles thereafter
Population: The study was stopped early for futility and EORTC QLQ Cancer Module (BR23) analysis was not performed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Capecitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib | Capecitabine
Serious Adverse Events (participants affected / at risk) | 72/238 | 44/240
Other Adverse Events (participants affected / at risk) | 228/238 | 229/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=238) | Capecitabine (N=240)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Diplopia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Disease progression (General disorders) | 14 | 8
Fatigue (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 3
Anal abscess (Infections and infestations) | 1 | 0
Fungal peritonitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=238) | Capecitabine (N=240)
Anaemia (Blood and lymphatic system disorders) | 23 | 22
Anisocytosis (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 19 | 13
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 43 | 28
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 38 | 5
Angina pectoris (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 1 | 3
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 6 | 4
Hyperthyroidism (Endocrine disorders) | 4 | 0
Hypothyroidism (Endocrine disorders) | 31 | 2
Thyroiditis chronic (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 7 | 8
Diplopia (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 3 | 3
Eye discharge (Eye disorders) | 2 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 2
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 8 | 1
Eyelid ptosis (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 7 | 9
Ocular surface disease (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 2 | 0
Pupils unequal (Eye disorders) | 0 | 1
Scleral pigmentation (Eye disorders) | 1 | 0
Scotoma (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 3 | 1
Visual impairment (Eye disorders) | 2 | 0
Xerophthalmia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 13 | 6
Abdominal pain (Gastrointestinal disorders) | 21 | 26
Abdominal pain lower (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 29 | 21
Abdominal rigidity (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 2 | 1
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 5 | 2
Cheilitis (Gastrointestinal disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 38 | 23
Dental caries (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 97 | 95
Dry mouth (Gastrointestinal disorders) | 18 | 10
Duodenitis (Gastrointestinal disorders) | 1 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 34 | 13
Dysphagia (Gastrointestinal disorders) | 6 | 5
Epigastric discomfort (Gastrointestinal disorders) | 4 | 2
Eructation (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 5 | 5
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 12 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Gingival bleeding (Gastrointestinal disorders) | 15 | 1
Gingival disorder (Gastrointestinal disorders) | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 8 | 0
Gingival swelling (Gastrointestinal disorders) | 3 | 1
Gingivitis (Gastrointestinal disorders) | 6 | 4
Glossitis (Gastrointestinal disorders) | 2 | 0
Glossodynia (Gastrointestinal disorders) | 5 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 4
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip discolouration (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 4 | 0
Mouth ulceration (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 94 | 75
Odynophagia (Gastrointestinal disorders) | 2 | 1
Oesophageal pain (Gastrointestinal disorders) | 1 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 3
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 5 | 1
Painful defaecation (Gastrointestinal disorders) | 2 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 3 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 39 | 22
Tongue ulceration (Gastrointestinal disorders) | 1 | 1
Tooth discolouration (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 88 | 34
Administration site pain (General disorders) | 0 | 1
Asthenia (General disorders) | 49 | 39
Axillary pain (General disorders) | 3 | 2
Chest discomfort (General disorders) | 1 | 3
Chest pain (General disorders) | 9 | 16
Chills (General disorders) | 4 | 2
Disease progression (General disorders) | 1 | 0
Extravasation (General disorders) | 0 | 1
Face oedema (General disorders) | 17 | 0
Fatigue (General disorders) | 82 | 61
Feeling hot (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 4
Generalised oedema (General disorders) | 4 | 0
Hyperthermia (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 2 | 0
Local swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Malaise (General disorders) | 7 | 4
Mucosal dryness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 59 | 36
Nodule (General disorders) | 0 | 1
Oedema (General disorders) | 10 | 2
Oedema peripheral (General disorders) | 19 | 21
Pain (General disorders) | 6 | 8
Pyrexia (General disorders) | 24 | 23
Sensation of foreign body (General disorders) | 0 | 1
Xerosis (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 5
Jaundice (Hepatobiliary disorders) | 2 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Iodine allergy (Immune system disorders) | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Breast infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2
Candidiasis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 3
Cystitis (Infections and infestations) | 2 | 2
Dacryocystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 3
Herpes zoster (Infections and infestations) | 2 | 1
Hordeolum (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 3 | 7
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nail infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 15 | 15
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 3
Oral herpes (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 4
Pharyngitis (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 4 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Urinary tract infection (Infections and infestations) | 12 | 4
Vaginal infection (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Vulvovaginitis (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 14 | 5
Aspartate aminotransferase (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 15 | 6
Blood albumin decreased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 2 | 6
Blood cholesterol decreased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 3 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 2 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 3 | 0
Blood thyroid stimulating hormone increased (Investigations) | 12 | 0
Blood urea increased (Investigations) | 2 | 0
Blood uric acid increased (Investigations) | 2 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 6 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Haemoglobin (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 5 | 7
Heart rate increased (Investigations) | 1 | 0
Heart sounds abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Leucine aminopeptidase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 2
Neutrophil count decreased (Investigations) | 16 | 6
Platelet count decreased (Investigations) | 27 | 3
Protein total decreased (Investigations) | 1 | 0
Prothrombin time shortened (Investigations) | 1 | 0
Pulmonary physical examination abnormal (Investigations) | 0 | 1
Thyroxine increased (Investigations) | 2 | 1
Transaminases increased (Investigations) | 2 | 0
Tri-iodothyronine free increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 10 | 10
Weight increased (Investigations) | 2 | 3
White blood cell count (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 15 | 12
Decreased appetite (Metabolism and nutrition disorders) | 67 | 48
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 18
Bone fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 21
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Ageusia (Nervous system disorders) | 6 | 0
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 10 | 15
Dizziness postural (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 61 | 11
Headache (Nervous system disorders) | 38 | 23
Hyperaesthesia (Nervous system disorders) | 1 | 1
Hyperreflexia (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 8 | 10
Lethargy (Nervous system disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 5
Nystagmus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 10
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 3
Polyneuropathy (Nervous system disorders) | 2 | 3
Sciatica (Nervous system disorders) | 3 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
VIth nerve disorder (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 7 | 5
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 5 | 7
Disorientation (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 21 | 14
Mood swings (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Perinephric effusion (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 9 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 2 | 1
Breast pain (Reproductive system and breast disorders) | 4 | 6
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 18
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 25
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 5 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 6
Blister (Skin and subcutaneous tissue disorders) | 1 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 13
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 7 | 5
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 8 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5 | 1
Koilonychia (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 2
Nail pigmentation (Skin and subcutaneous tissue disorders) | 3 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 80 | 149
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 28 | 19
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 18 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 23
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 5
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 4 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 19 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 5 | 0
Haemorrhage (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 4 | 5
Hypertension (Vascular disorders) | 53 | 6
Hypotension (Vascular disorders) | 1 | 2
Lymphoedema (Vascular disorders) | 3 | 7
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to patient enrollment termination, PFS/OR/TTP/DR were done by investigator assessment due to lack of central review data and TTR/EORTC QLQ-C30/QLQ BR23 analyses were not done. Those enrolled could receive capecitabine or enter an extension trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.